CLINICAL TRIAL: NCT06175234
Title: A Study Evaluating the User Experience With the FARAVIEW™ Technology of the RHYTHMIA HDx™ Mapping System When Used With the FARAWAVE NAV™ Pulsed Field Ablation Catheter in the Treatment of Atrial Fibrillation
Brief Title: Feasibility Study on the FARAVIEW Technology
Acronym: NAVIGATE PF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PF305
Record Dates: First submitted 2023-11-27; First posted 2023-12-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter ablation for Paroxysmal or Persistent Atrial Fibrillation (Other): Subjects scheduled to undergo endocardial mapping and Pulmonary Vein Isolation (PVI) in the treatment of atrial fibrillation. For patients with persistent AF, left atrial posterior wall isolation (PWI) may also be performed in addition to PVI at the discretion of the investigator
  Interventions: Device: Ablation Treatment

INTERVENTIONS:
Device: Ablation Treatment — For subjects with paroxysmal AF, Pulmonary Vein Isolation will be performed with the FARAWAVE NAV catheter. For subjects with persistent AF, left atrial posterior wall isolation (PWI) may also be performed at the discretion of the investigator, with the FARAWAVE NAV PFA catheter.

SUMMARY:
The purpose of this study is to gather data regarding the utilization of the FARAVIEW™ feature of the RHYTHMIA HDx Mapping System when used in conjunction with the FARAWAVE NAV Pulsed Field Ablation catheter in subjects undergoing catheter-based endocardial mapping and catheter-based ablation treatment of Atrial Fibrillation.

DETAILED DESCRIPTION:
The objective of this study is to obtain First-in-Human (FIH) experience with the FARAVIEW™ technology of the RHYTHMIA HDx™ Mapping System when it is used to visualize and track the FARAWAVE NAV™ Pulsed Field Ablation (PFA) catheter in the treatment of Atrial Fibrillation (AF). The study will collect FIH data on user experience and workflow using the FARAVIEW technology to visualize and track the FARAWAVE NAV PFA catheter (part of the FARAPULSE™ Pulsed Field Ablation System). Subjects with Paroxysmal and Persistent Atrial Fibrillation will be included in this study.

NAVIGATE PF Phase 2 has the same objective of the NAVIGATE PF study and incorporates a Day 60 remapping procedure and Day 90 safety follow-up. This procedure has the additional objective to assess durability of isolation and to compare electro-anatomical maps information between Index procedure and Day 60 remapping. One clinical site in Europe that participated in NAVIGATE PF and enrolled under protocol ver A., will contribute enrollments in Phase 2 of the NAVIGATE PF study. Approximately 30 subjects will be enrolled in Phase 2 of the NAVIGATE PF study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years of age, or older if required by local law
2. Symptomatic, documented, drug-resistant, Atrial Fibrillation

   1. Documented: at a minimum a physician's note confirming the arrhythmia symptoms and durations AND within 180 days of the Enrollment Date one (1) ECG from any regulatory cleared rhythm monitoring device showing AF
   2. Drug-resistant: effectiveness failure of, intolerance to, or specific contraindication to at least one (1) AAD (Class I, II, III or IV) 1
3. Informed consent: willing and capable of providing informed consent
4. Full participation: willing and capable of participating in all follow-up assessments and testing associated with this clinical investigation at an approved clinical investigational center

Exclusion Criteria:

1. Atrial exclusions - Any of the following atrial conditions:

   1. Prior atrial ablation: any prior atrial endocardial, epicardial or surgical ablation procedure for arrhythmia other than ablation for right sided SVT or cavotricuspid isthmus ablation
   2. Atrial myxoma: current atrial myxoma
   3. Pulmonary veins: any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
   4. Atrial thrombus: current left atrial thrombus
   5. Long standing persistent AF: continuous AF lasting longer than 12 months
2. Cardiovascular exclusions - Any of the following CV conditions:

   1. Ventricular arrhythmia: history of sustained ventricular tachycardia or any ventricular fibrillation
   2. Secondary AF: AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
   3. Cardiac devices and implants: current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, interatrial baffle, closure device, patch, or patent foramen ovale or ASD occluder, LA appendage closure, device or occlusion.
   4. Clinically significant valvular disease: valvular disease that is any of the following:

   i. Symptomatic ii. Causing or exacerbating congestive heart failure iii. Associated with abnormal LV function or hemodynamic measurements e. Cardiomyopathy i. Hypertrophic cardiomyopathy ii. Cardiac amyloidosis f. Valve prostheses: any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty g. Access issues: any IVC filter, known inability to obtain vascular access or other contraindication to femoral access h. Rheumatic disease: rheumatic heart disease i. Anticipated cardiac surgery: awaiting cardiac transplantation or other cardiac surgery within the next 12 months
3. Any of the following conditions at baseline (Section 10.4):

   1. Heart failure NYHA Heart failure associated with NYHA IV
   2. Ejection fraction: LVEF < 40%
4. Any of the following events within 90 Days of the Consent Date:

   1. Coronary disease: myocardial infarction (MI), unstable or coronary intervention
   2. Cardiac surgery: any cardiac surgery
   3. Heart failure hospitalization: heart failure hospitalization
   4. Pericardium: pericarditis or symptomatic pericardial effusion
   5. GI bleeding: gastrointestinal bleeding
   6. Neurovascular event: stroke, TIA, or intracranial bleeding
   7. Thromboembolism: any non-neurologic thromboembolic event
   8. Carotid intervention: carotid stenting or endarterectomy
5. Bleeding diathesis: thrombocytosis, thrombocytopenia, disorder of blood clotting or bleeding diathesis
6. Contraindication to anticoagulation: contraindication to, or unwillingness to use, systemic anticoagulation
7. Pregnancy: women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
8. Health conditions that in the investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:

   1. Obesity: Body Mass Index (BMI) > 45.0
   2. Transplantation: solid organ or hematologic transplant, or currently being evaluated for a transplant
   3. Diaphragmatic abnormality: any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
   4. Pulmonary: severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
   5. Renal: renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
   6. Malignancy: active malignancy (other than cutaneous basal cell or squamous cell carcinoma)
   7. Gastrointestinal: clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
   8. Infections: active systemic infection
   9. COVID-19 disease: known positive test for COVID-19 and disease not clinically resolved
9. Life expectancy: predicted life expectancy less than one (1) year
10. Participation in another trial: subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility
11. Congenital heart disease: congenital heart disease with any clinically significant residual anatomic or conduction abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with PVI success | At the end of the ablation procedure
  PVI success is defined as the proportion of veins isolated vs reconnected at the end of the procedure as assessed by a site's standard of care method for testing vein isolation
Number of subjects with PWI success | At the end of the ablation procedure
  PWI success is defined as the isolation of the left atrial PW at the end of the procedure as assessed by a site's standard of care method for testing
Physician feedback on FARAVIEW technology of the RHYTHMIA mapping system by means of a questionnaire | At the end of the ablation procedure
  Physician feedback on the FARAVIEW technology of the RHYTHMIA mapping system will be collected by means of a questionnaire.
umber of subjects presenting with PV or PW reconnections site's standard of care method. Procedural complications: device and/or procedure-related AEs. | At the end of the ablation procedure
  Device and/or procedure-related AEs will be collected to evaluate the procedural complications rate.

OTHER OUTCOMES:
Number of subjects presenting with PV or PW reconnections (NAVIGATE PF Phase 2 only) | Day-60 remapping procedure
  Number of subjects presenting with PV or PW reconnections at the Day-60 remapping procedure, as assessed by a site's standard of care method.
Comparison of electro-anatomical maps (NAVIGATE PF Phase 2 only) | Day-60 remapping procedure
  Comparison of electro-anatomical maps Index Procedure vs Day 60

CONTACTS AND LOCATIONS:
Locations (3):
- Na Homolce Hospital, Prague, Czechia
- Mater Private Hospital, Dublin, Ireland
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Garcia-Bolao I, Reddy VY, Su WW, Koruth JS, Fitzpatrick N, Neuzil P, Rincon RA, Canepa S, Kang K, Oesterlein T, Koop BE, Metzdorff C, Okeson B, Gutbrod SR, Szeplaki G. Visualization of PFA During PVI With the Second-Generation Pentaspline Catheter: NAVIGATE-PF Phase 1 Results. JACC Clin Electrophysiol. 2025 Dec 30:S2405-500X(25)00998-3. doi: 10.1016/j.jacep.2025.11.016. Online ahead of print. PMID 41474406